CLINICAL TRIAL: NCT01439932
Title: Effectiveness of Manual Therapy Combined With Standard Treatment in the Management of Plantar Fasciitis, a Randomized Control Trial
Brief Title: Effectiveness of Manual Therapy Combined With Standard Treatment in the Management of Plantar Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Collaborators: Clalit Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: MMC11XXX-XXKCTIL; PF-001-ISR (Other: Clalit Health Services)
Record Dates: First submitted 2011-09-20; First posted 2011-09-23 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2011-09

CONDITIONS: Plantar Calcaneal Spur; Fasciitis, Plantar
Keywords: plantar fasciitis; heel pain; manual treatment; dorsi flexion
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- ankle mobilization for pain release (Experimental): stretching exercise for the plantar fascia and triceps surae muscles three times a day throughout the study period.
  During each visit the exercise performance will be checked by the therapist. In addition, participants from both groups will get ultra sound therapy in frequency of 1 MHz, power of 1.5 watts per centimeter-squared, pulses of 50% for 5 minutes.
  The study group will receive the same treatment and a number of manual techniques that include antero-posterior (AP) mobilization for talocrural joint in two variations (weight baring and non-weight baring) to improve the range of dorsi flexion, subtalar joint mobilization to improve range of eversion and mid-tarsal mobilization to improve pronation / supination of the forefoot. Each technique will be carried out for 1 to 1.5 minutes for a total of 5 minutes of manual treatment.
  All patients will receive information and guidance to practice at home.
  Interventions: Device: algometer

INTERVENTIONS:
Device: algometer — Pressure algometer (Algometry) - This is an instrument that measures pain threshold (the minimum pressure required to produce pain). The instrument consists of a flat disk size centimeter square attached to pressure transducer and measuring electrodes. The disk is placed vertically on the point of pain and therapist increases the intensity of the pressure until initial pain appears (when sense of pressure becomes sense of pain.) Score is determined by average of three repeated measurements with 30 seconds break between each.
  The algometer allows an objective assessment of pain in addition to LEFS score which is a subjective tool. The algometer test was found to be valid and reliable in repeated measurements (interrater, intrarater) by Andrew A. Fischerin 1987 with healthy people [Andrew 1987]. In another study high reliability was found for averaging between three repeated tests: ICC = 0.91 (CI 0.82; 0.97 95%). [Linda et al 2007]
  Other Names: SBMEDIC Electronics

SUMMARY:
Background: Plantar fasciitis (PF) is a common problem that tends to attack about 10% of the population during life. This is a degenerative condition of the plantar fascia at its insertion at the bottom of the heel. Pain appears mainly on the first steps in the morning or after prolonged lack of weight bearing. The pain intensity can be very high and this can cause functional limitations and reduce quality of life.

Despite the high prevalence of the PF, treatment is controversial and not supported by extensive research. Review of the previous studies on various treatments, mentioned steroid injections, shock waves, night splint, orthotics, heel padding and stretching exercises.

Limitation of ankle dorsi flexion is a common finding and thought to be a contributing factor to the development of pathology. So far, this issue had been addressed mainly by soft tissue therapy techniques to improve ankle range of motion in patients with PF. Only one study (Joshua et al 2009) evaluated the effect of ankle joint mobilizations of PF. However, in this study mobilizations were part of complex therapy and therefore the effect of treatment cannot be attributed solely to them.

The purpose of this study is to evaluate the effectiveness of ankle and mid-foot joints mobilization on pain and function of patients with PF.

The hypothesis is that manual mobilizations of ankle and midfoot joints in addition to conventional physical therapy will improve pain and function significantly more than conventional treatment, in patients with PF.

Methods: 50 patients, age 18-75 with a diagnosis of PF that meet the inclusion criteria will be recruited and randomly divided into two groups. Both groups will receive commonly accepted physical therapy treatment that includes stretching exercise of the plantar fascia and triceps surae muscles and ultrasound therapy at the site of symptoms. The study group will receive in addition manual mobilizations to the ankle and midfoot joints. The procedures will take place at the physiotherapy clinic Bat-Yamon of General Health Services and will last four weeks, twice a week.

DETAILED DESCRIPTION:
A prospective randomized double-blinded controlled clinical trial. Setting: Bat-Yamon physical therapy clinic of Clalit health services in Bat Yam.

Ethical considerations: The research proposal will be submitted for the approval of the Helsinki Committee at Meir Hospital in Kefar Saba. All patients will sign informed consent form according to the laws of medical ethics.

Subjects will be recruited from all the population of patients who are referred to physical therapy for the treatment of PF with diagnosis of plantar fasciitis or calcaneal spur.

Randomization will be carried out using envelopes that will be prepared in advance. Each patient will receive at the end of the baseline examination envelope with the type of treatment for which will be delivered only to the therapist so that the examiner and the patient will be blind to the treatment group.

Baseline and final evaluations will be performed by the examiner-therapist and treatments performed by three physical therapists at the Bat-Yamon clinic with experience of at least 3 years which will receive proper instruction and training.

Baseline examination will be performed after completing informed consent form and will include demographic information to be filled by patient, clinical interview and examination by the examiner. Demographic information includes age, gender, weight, BMI (calculated by the examiner), history of the problem, habits related to physical activity and occupation and general health.

The interview will refer to etiology and nature of symptoms. The clinical examination will include observation of foot structure and gait pattern, the presence of hit or swelling. Palpation for pain location and for ruling out fat pad Syndrome, clunk test and neurodynamic of tibial nerve will be performed to rule out tarsal tunnel syndrome (TTS). Patients with suspicion for one of these diagnoses will not be recruited. Dorsi flexion range of motion in both legs will be measured and compared to the range at the end of treatment. Measurement will be taken in two ways, once weight bearing with inclinometer - the patient stands in lounge position while tested leg in front and asked to bend the knee of this leg as possible without lifting the heel off the floor. The angle measured is the angle between the tibia and a vertical line to the floor.Second time without weight bearing with Goniometer- the patient lies on his back with a pillow under the tested knee , the therapist performs maximum dorsi flexion passively and asks the patient to add an active movement in the same direction. The angle measured is between fibula and fifth metatarsus

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75
* Pain allocated at the bottom of heel and produced by pressure
* Pain in the morning at first steps or after prolonged non-weight bearing
* NPRS morning pain score of 3 or higher

Exclusion Criteria:

* Tumors
* Prolonged use of steroids
* Fracture below knee during the last year
* Prior foot surgeries
* A positive diagnosis of Tarsal Tunnel Syndrome (TTS) / Fat Pad Syndrome
* Pregnancy
* Lack of availability in the coming month

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-10; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale 0-10 | one year and two months
  The participant will rate his pain intensity at first step in the morning on a scale of numbers between 0-10 when 0 means "no pain" and 10 means "very severe pain". NPRS is a valid and reliable tool for assessment of pain intensity and is a common tool in studies on PF.

CONTACTS AND LOCATIONS:
Overall Officials: Anat Shashua, BPT, Study Director
Locations (1):
- Clalit Health Services, Tel-Aviv district, Bat Yamon, Bat Yam, Israel

REFERENCES:
- [Derived] Shashua A, Flechter S, Avidan L, Ofir D, Melayev A, Kalichman L. The effect of additional ankle and midfoot mobilizations on plantar fasciitis: a randomized controlled trial. J Orthop Sports Phys Ther. 2015 Apr;45(4):265-72. doi: 10.2519/jospt.2015.5155. Epub 2015 Mar 4. PMID 25739844